CLINICAL TRIAL: NCT01508611
Title: Cost-efficacy of Silver Diammine Fluoride to Control Caries Lesions in Erupting Permanent First Molars - Randomized Clinical Trial.
Brief Title: Cost-efficacy of Silver Diammine Fluoride in Erupting Molars
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: University of Sao Paulo (Other)
Responsible Party: Principal Investigator, Mariana Minatel Braga, PhD, Associate Professor, University of Sao Paulo
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: SDFtrials-02
Record Dates: First submitted 2011-12-20; First posted 2012-01-12 (Estimated); Last update posted 2018-03-21 (Actual); Status verified 2018-03

CONDITIONS: Dental Caries
Keywords: dental caries; permanent teeth; silver diamine fluoride; tooth eruption
MeSH Terms: conditions — Dental Caries; Exanthema | interventions — silver diamine fluoride; Oral Hygiene

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 30% silver diammine fluoride (Active Comparator): The 30% silver diamine fluoride (Cariestop, Biodinamica) will be applied in erupting molars with a disposable microbrush for 3m. Then the surface will be washed for 30s.
  Interventions: Other: 30% silver diammine fluoride
- cross-toothbrushing (Active Comparator): Children will be oriented to proceed cross-toothbrushing in erupting molars
  Interventions: Behavioral: Oral hygiene

INTERVENTIONS:
Other: 30% silver diammine fluoride — The 30% silver diamine fluoride (Cariestop, Biodinamica) will be applied with a disposable microbrush for 3m. Then the surface will be washed for 30s.
  Anteroposterior toothbrushing technique will be explained to the children.
  Other Names: Cariestop; Biodinamica
  Arms: 30% silver diammine fluoride
Behavioral: Oral hygiene — With the patient's own brush, supervised brushing the erupting molar with fluoridated toothpaste will be guided using the cross-toothbrushing technique
  Other Names: Toothbrush
  Arms: cross-toothbrushing

SUMMARY:
This study aims to evaluate the cost-effectiveness of 30% silver diammine fluoride in the treatment of clinically caries lesions in enamel, on occlusal surfaces in first permanent molars compared to a control group that performs only the cross-toothbrushing technique and evaluate the acceptability and satisfaction of patients and responsible for the application of the solution cariostatic.

DETAILED DESCRIPTION:
The sample will be comprised of 183 patients between 4 to 7 year-old, who present at least occlusal surface with initial caries lesion (ICDAS 1, 2, 3). Patients will be randomly allocated to treatments, according to the technique to be employed: (I) 30% diamine silver fluoride, (II) cross-toothbrushing technique. Will also be guided and motivated individual, where these children will be taught the technique of brushing conventional. It will be given to all patients a toothbrush. In times of reassessment, the degree of wear of the bristles of these brushes will be evaluated in order to infer the use of the same. The teeth will be evaluated by clinical and exams at baseline and after 3, 6, 12, 18 and 24 months.

ELIGIBILITY:
Inclusion Criteria:

* erupting permanent molars (that are not in full occlusion)
* not special children
* children who present at least occlusal surface with initial caries lesion (ICDAS 1, 2, 3)

Exclusion Criteria:

* presence of cavitated caries lesions
* presence of enamel defects (hypoplasias)

Ages: 4 Years to 7 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 192 (Actual)
Dates: Start 2015-02; Primary Completion 2018-08 (Estimated); Study Completion 2019-08 (Estimated)

PRIMARY OUTCOMES:
Caries progression | 12 months

SECONDARY OUTCOMES:
cost | 24 months
patient's satisfaction | 24 months
patient's discomfort | 24 months
duration | 24 months

CONTACTS AND LOCATIONS:
Overall Officials: Mariana M Braga, PhD, Principal Investigator — USao Paulo
Locations (1):
- Universidade de Sao Paulo, São Paulo, Brazil

REFERENCES:
- [Background] Braga MM, Mendes FM, De Benedetto MS, Imparato JC. Effect of silver diammine fluoride on incipient caries lesions in erupting permanent first molars: a pilot study. J Dent Child (Chic). 2009 Jan-Apr;76(1):28-33. PMID 19341576
- [Background] Chu CH, Lo EC, Lin HC. Effectiveness of silver diamine fluoride and sodium fluoride varnish in arresting dentin caries in Chinese pre-school children. J Dent Res. 2002 Nov;81(11):767-70. doi: 10.1177/0810767. PMID 12407092
- [Background] Ekstrand KR, Martignon S, Ricketts DJ, Qvist V. Detection and activity assessment of primary coronal caries lesions: a methodologic study. Oper Dent. 2007 May-Jun;32(3):225-35. doi: 10.2341/06-63. PMID 17555173
- [Background] Ekstrand KR, Ricketts DN, Kidd EA, Qvist V, Schou S. Detection, diagnosing, monitoring and logical treatment of occlusal caries in relation to lesion activity and severity: an in vivo examination with histological validation. Caries Res. 1998;32(4):247-54. doi: 10.1159/000016460. PMID 9643366
- [Background] Ismail AI, Sohn W, Tellez M, Amaya A, Sen A, Hasson H, Pitts NB. The International Caries Detection and Assessment System (ICDAS): an integrated system for measuring dental caries. Community Dent Oral Epidemiol. 2007 Jun;35(3):170-8. doi: 10.1111/j.1600-0528.2007.00347.x. PMID 17518963
- [Background] Llodra JC, Rodriguez A, Ferrer B, Menardia V, Ramos T, Morato M. Efficacy of silver diamine fluoride for caries reduction in primary teeth and first permanent molars of schoolchildren: 36-month clinical trial. J Dent Res. 2005 Aug;84(8):721-4. doi: 10.1177/154405910508400807. PMID 16040729
- [Background] Yee R, Holmgren C, Mulder J, Lama D, Walker D, van Palenstein Helderman W. Efficacy of silver diamine fluoride for Arresting Caries Treatment. J Dent Res. 2009 Jul;88(7):644-7. doi: 10.1177/0022034509338671. PMID 19641152